CLINICAL TRIAL: NCT00599443
Title: Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Tolerability of a Cell-Derived Influenza Vaccine in Healthy Adults Aged ≥18 Years and ≤ 49 Years.
Brief Title: Safety and Tolerability of a Cell-Derived Influenza Vaccine in Healthy Adults Aged ≥18 Years and ≤ 49 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Wil Cramer, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S203.1.001
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: Cell-derived subunit influenza vaccine; Safety; Reactogenicity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Seasonal cell-derived influenza vaccine
- 2 (Placebo Comparator)
  Interventions: Biological: Placebo Comparator

INTERVENTIONS:
Biological: Seasonal cell-derived influenza vaccine — 0.5 mL im, single dose
  Arms: 1
Biological: Placebo Comparator — 0.5 mL im, single dose
  Arms: 2

SUMMARY:
A controlled, double blinded study to determine the safety and reactogenicity in healthy adults of a single dose of a trivalent cell-derived influenza vaccine administered by intramuscular injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female or male subjects aged ≧18 and ≦49 years
* Willing and able to give informed consent

Exclusion Criteria:

* Influenza vaccination of laboratory confirmed influenza infection within six months of informed consent,
* presence of any significant medical condition,
* a serious adverse reaction after a previous (influenza) vaccination,
* underlying medical conditions for which annual influenza vaccine is recommended by the Advisory Committee on Immunization Practices (ACIP),
* chronic diseases requiring long-term immunosuppressive therapy

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of one dose of cell-derived influenza vaccine in healthy adults aged ≧18 years and ≦ 49 years after vaccination. | 3 weeks
Long-term safety | 6 months

SECONDARY OUTCOMES:
HI antibody titers | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals